CLINICAL TRIAL: NCT02717936
Title: Prospektive Therapie-Studie Zur Behandlung Des Desmoplastischen Plattenepithelkarzinoms
Brief Title: Investigation of Desmoplastic Squamous Cell Carcinoma
Acronym: DesmoPEK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DESMOPEK1
Record Dates: First submitted 2016-01-27; First posted 2016-03-24 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-01

CONDITIONS: Squamous Cell Carcinoma of the Skin
Keywords: squamous cell carcinoma; dermatosurgery; immunohistochemistry
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Immunohistochemistry (Other): Patients are investigated using immunohistochemistry with Pancytokeratin
  Interventions: Procedure: Immunohistochemistry using Pancytokeratin Staining

INTERVENTIONS:
Procedure: Immunohistochemistry using Pancytokeratin Staining

SUMMARY:
Aim of the study is to verify wether it is possible to have a more sensitive diagnostic tool using pancytokeratin immunohistochemistry for desmoplastic squamous cell carcinoma compared to regular H&E staining. The investigators therefore plan to include 73 participants with a confirmed diagnosis of desmoplastic squamous cell carcinoma and do regular follow up.

ELIGIBILITY:
Inclusion Criteria:

* desmoplastic squamous cell carcinoma (SCC) of the skin

Exclusion Criteria:

* tumor recurrence
* collision tumors
* other skin malignancies
* progeria
* Rothmund-Thomson-Syndrome
* lacking of the capacity for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival of patients with desmoplastic squamous cell carcinoma (SCC) diagnosed with immunohistochemistry . | 4 years

SECONDARY OUTCOMES:
Reduction of local recurrence with immunohistochemistry | 4 years
Histological pattern of tumour growth (continuous versus discontinuous) | 4 years
Dimension of the tumor spreading according to histological work-up (measured in mm) | 4 years
Presence of perineurial and perivascular tumor invasion according to histological work-up | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Universityhospital, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided